CLINICAL TRIAL: NCT02998385
Title: A Phase III Randomized Study of Chemo-radiotherapy Versus Radiotherapy Alone in the Adjuvant Treatment of Salivary Glands and Nasal Tumors (IMRT or Protontherapy)
Brief Title: Chemo-radiotherapy Versus Radiotherapy in the Treatment of Salivary Glands and Nasal Tumors (IMRT or Protontherapy)
Acronym: SANTAL
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Groupe Oncologie Radiotherapie Tete et Cou (Other)
Collaborators: National Cancer Institute, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GORTEC 2016-02
Record Dates: First submitted 2016-12-15; First posted 2016-12-20 (Estimated); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: HNSCC
Keywords: salivary glands; sinus carcinoma; radiochemotherapy concomitant; cisplatin; protontherapy
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck | interventions — Cisplatin; Radiotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Radiotherapy (Active Comparator): Arm A
  Radiation therapy: 66 to 70 Gy in fractions of 2 Gy, 1 fraction/day, 5 fractions per week.
  Radiation therapy will be conducted by conformational intensity modulation radiotherapy (IMRT) or protontherapy. Irradiation by 3D conformational radiotherapy can be discussed on a case by case with the Intergroup Coordinator GORTEC.
  Interventions: Radiation: radiotherapy
- Radiotherapy + concomitant cisplatin (Experimental): Arm B Concomitant systemic treatment with cisplatin + radiotherapy
  According to standard protocol of concomitant cisplatin 100 mg/m2 IV on day 1 - J22 - 43 (3 maximum cycles).
  Radiation therapy: 66 to 70 Gy in fractions of 2 Gy, 1 fraction/day, 5 fractions per week.
  Radiation therapy will be conducted by conformational intensity modulation radiotherapy (IMRT) or protontherapy. Irradiation by 3D conformational radiotherapy can be discussed on a case by case with the Intergroup Coordinator GORTEC
  Interventions: Drug: Cisplatin; Radiation: radiotherapy

INTERVENTIONS:
Drug: Cisplatin — intravenous, concomitant to irradiation
  Arms: Radiotherapy + concomitant cisplatin
Radiation: radiotherapy — 66 à 70 Gy per fractions of 2 Gy, 1 fraction/day, 5 fractions/week

SUMMARY:
A phase III, multicenter, randomized, open-label, french study comparing:

* Arm A : Radiotherapy alone (66 to 70 Gy; 5 fractions/week; 1fraction/day; 2 Gy/fraction) (IMRT or protontherapy)
* Arm B: Radiotherapy (66 to 70 Gy; 5 fractions/week; 1fraction/day; 2 Gy/fraction; IMRT or protontherapy) + concomitant cisplatin 100 mg/m2 IV on day 1 - J22 - 43 (3 cycles)

DETAILED DESCRIPTION:
Carcinomas of the sinuses and the salivary glands are rare. They are heterogeneous in terms of anatomical sites and histology subtypes. For this reason and in the absence of prospective study, their treatment is still largely extrapolated from data of frequent carcinomas of the upper digestive tract. These tumors are most often diagnosed lately. Their treatment is based on a multimodal management of care, with a central place for the surgery and radiotherapy (Proof level Grade C). Despite the advances in surgical techniques, and the addition of radiation therapy, the 5-year overall survival probability does not exceed 65% mainly due to a loco regional development.

In this context, a chemotherapy administered concomitantly to radiotherapy, could increase the efficacy of the locoregional treatment by a radiosensibilization process and regardless of the histology. This point is regularly discussed in multidisciplinary concertation meeting, including bi-monthly national REFCOR meeting (network of French Expertise on rare Cancers of the head and neck). At present, the lack of data brings even to discuss the addition of cisplatin to exclusive irradiation of unresectable or not operable tumors.

No randomized study has been published in this context. The first comparative prospective study addressing the addition of weekly cisplatin to the adjuvant irradiation of salivary, is a phase II randomized study (Radiation Therapy Oncology Group - RTOG 1008) currently enrolling patients in the United States of America.

The Sponsor propose to conduct a phase III randomized study evaluating the impact of the addition of cisplatin to a treatment by radiotherapy in adjuvant setting (≥ 65 Gy) in case of a high risk of recurrence: case of radioresistant histologies (e.g. cystic fibrosis adenoids carcinomas), or case of unfavourable histo-prognostic criteria (incomplete resection, presence of emboli, etc.) in this population.

ELIGIBILITY:
Inclusion Criteria:

- Resected tumors of the sinus or the salivary glands T3-4, N1-3 or T1-2 N0, with overgrown banks or positive margins (< 5 mm)

or

Unresectable or not operable tumors of salivary glands or sinuses

* Carcinomas of the main salivary glands (parotid, submandibular or sublingual glands) and accessories or Malignant sinus tumors with any histological type except melanoma, lymphoma, mesenchymal tumor (sarcoma type), squamous cell carcinoma and nasopharyngeal carcinoma type 1, 2, 3.
* Age ≥ 18 years
* Performance status 0 -2 (WHO criteria)
* For patients ≥ 70 years, the score to the G8 questionnaire must be > 14 with no fall in the previous 12 months or with a geriatric assessment consistent with the administration of chemotherapy
* Estimated life expectancy greater than or equal to 6 months
* Neutrophils > 1.5 x 109/l, platelets > 100 x 109/l, hemoglobin ≥ 9.5 g/dl, bilirubin ≤ 3 x upper normal value (ULN), AST/ALT < 5 ULN, PAL < 3 ULN
* Creatinin Clearance ≥ 60 mL/min (Cockroft formula)
* Adequate cardiac function according to the investigator, compatible with the administration of cisplatin 100 mg/m²
* Affiliation to a social insurance or beneficiary of such a regimen
* Patient having given his written consent signed before any study specific procedure.

Exclusion Criteria:

* History of radiotherapy in the ENT region and/or neoadjuvant chemotherapy for the pathology concerned
* Synchronous metastases
* Contraindications for administration of cisplatin or carboplatin
* Allergy to cisplatin and/or its excipients
* Vaccination against yellow fever, recent or planned
* Administration of phenytoin with prophylactic purpose
* Other cancer, except for cancer in situ of the cervix, skin Carcinoma (except melanoma) or cancer controlled for more than 5 years
* Pregnant, breastfeeding or without birth control woman. Woman having the ability to procreate should have (serum or urinary) negative pregnancy test within 14 days prior to study treatment decision-making. (Men or women) patients should use a reliable contraceptive method throughout the treatment and at least 6 months after the end of chemotherapy.
* Persons deprived of liberty under supervision or under curatorship, or unable to adhere to medical follow-up of the study for geographical, social or psychological reasons.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 342 (Estimated)
Dates: Start 2017-01-20 (Actual); Primary Completion 2030-02 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | From date of randomization to date of disease progression or death, which occur first, assessed during 62 months
  Compare progression-free survival between the 2 treatment arms: radiation therapy alone versus radiochimiotherapy in adjuvant patients treatment operated.

SECONDARY OUTCOMES:
Overall Survival | From date of randomization to date of death, assessed during 62 months
  Compare the 2 arms of treatment in operated patients in terms of overall survival

OTHER OUTCOMES:
Assessment of quality of Life: QLQC30 overall score | From date of randomization to end of study or death or progression (the first occurred), assessed during 62 months
  Compare quality of life (QLQC30 overall score) between arms

CONTACTS AND LOCATIONS:
Locations (1):
- Hôpital Bégin, Saint-Mandé, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferrari M, Orlandi E, Bossi P. Sinonasal cancers treatments: state of the art. Curr Opin Oncol. 2021 May 1;33(3):196-205. doi: 10.1097/CCO.0000000000000726. PMID 33756515
- [Derived] Joshi NP, Broughman JR. Postoperative Management of Salivary Gland Tumors. Curr Treat Options Oncol. 2021 Feb 9;22(3):23. doi: 10.1007/s11864-021-00820-9. PMID 33560478